CLINICAL TRIAL: NCT02480738
Title: Effectiveness of Computerized Cognitive Training Apparatus (CoCoTA) in the Elderly With Normal Cognition, Subjective Cognitive Impairment, Mild Cognitive Impairment
Brief Title: Effectiveness of Computerized Cognitive Training in the Elderly With Cognitive Impairment
Acronym: CoCoTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, SangYun Kim, Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10035434
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Mild Cognitive Impairment
Keywords: subjective cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mild cognitive impairment (Experimental): Intervention: Computerized Cognitive Training Apparatus
  Interventions: Behavioral: Computerized Cognitive Training Apparatus
- Subjective cognitive impairment (Experimental): Intervention: Computerized Cognitive Training Apparatus
  Interventions: Behavioral: Computerized Cognitive Training Apparatus
- Normal controls (Active Comparator): Intervention: Computerized Cognitive Training Apparatus
  Interventions: Behavioral: Computerized Cognitive Training Apparatus

INTERVENTIONS:
Behavioral: Computerized Cognitive Training Apparatus — CoCoTA was developed through collaborative research with the Korean Institute of Science and Technology (KIST) and Primpo Co. Ltd. (www.primpo.com). It was designed to stimulate numerous cognitive domains simultaneously by using sounds and objects familiar to Korean elderly. Training themes and scenarios were developed and evaluated by six board-certified neurologists and three neuropsychologists who specialize in dementia.
  Each subject participated in a total of 24 sessions of cognitive training, which consisted of 40 minutes of training, twice per week. To assure the consistency of cognitive training, trained personnel stayed nearby the subjects to help throughout the training process.
  Other Names: CoCoTA

SUMMARY:
This study is to investigate the effectiveness of computerized cognitive training, and corresponding neural substrates through multimodal neuroimaging assessment, in the elderly with normal cognition, subjective cognitive impairment, and mild cognitive impairment.

DETAILED DESCRIPTION:
Computerized cognitive training has the advantage of easy accessibility for community-dwelling elderly. It can be much cheaper than traditional neuropsychological training methods, which require trained neuropsychologists. Furthermore, it may be more fun and easier to be optimized to an individual patients' cognitive status than other traditional methods.

Clinical efficacy of these kinds of cognitive training applications has been validated through several studies. A recent systematic review reported that the domains of working memory, executive function, and processing speed benefited the most by classic computerized cognitive training tasks, and that these benefits were comparable with traditional cognitive training methods. Apart from neuropsychological data, neuroimaging studies focusing on the effectiveness of computerized cognitive training are scant.

There have been no previous studies investigating the possible neural substrates of computerized cognitive training using multimodal neuroimaging modalities simultaneously. Thus, we aimed to investigate the effectiveness of computerized cognitive training and corresponding neural substrates in subjects with mild cognitive impairment, subjective memory impairment, and normal controls through a multimodal approach.

ELIGIBILITY:
Inclusion Criteria:

* Ages >50 to ≤70
* Years of education ≥ 6 years
* No physical barrier preventing the dominant hand from using the computer mouse

Exclusion Criteria:

* Subjects who had any structural lesions or psychiatric disorders that explained the memory deficits
* Subjects had to be able to undergo pre- and post-training evaluations such as electroencephalography (EEG), FDG-PET, and magnetic resonance imaging (MRI)
* Subjects who had scalp lesions, severe back pain, or claustrophobia that precluded pre- and post-training evaluations.

Ages: 51 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Clinical improvement in the follow-up neuropsychological tests | 12 weeks
  changes in memory and frontal domain subscores between the baseline and follow-up

SECONDARY OUTCOMES:
Cortical thickness changes between baseline and follow-up volumetric MRI | 12 weeks
  surface-based morphometry using freesurfer software
White matter integrities changes between baseline and follow-up diffusion tensor imaging | 12 weeks
  tract-based spatial statistics using fsl software
Spectral ratio changes between baseline and follow-up EEG | 12 weeks
  EEG spectral ratio analysis
local activation pattern changes between baseline and follow-up Fludeoxyglucose PET | 12 weeks
  local activation pattern analysis using SPM

CONTACTS AND LOCATIONS:
Overall Officials: SangYun Kim, MD,PhD, Principal Investigator — Seoul National University Bundang Hospital

REFERENCES:
- [Result] Na HR, Lim JS, Kim WJ, Jang JW, Baek MJ, Kim J, Park YH, Park SY, Kim S. Multimodal Assessment of Neural Substrates in Computerized Cognitive Training: A Preliminary Study. J Clin Neurol. 2018 Oct;14(4):454-463. doi: 10.3988/jcn.2018.14.4.454. Epub 2018 Jun 26. PMID 30198220